CLINICAL TRIAL: NCT05817071
Title: Results of Arthroscopic Massive Rotator Cuff Tears Repair With Or Without Superior Capsular Augmentation Using Proximal Part Of Long Head Of Biceps Tendon: A Randomized Controlled Trial
Brief Title: Results of Arthroscopic Massive Rotator Cuff Tears Repair With or Without Using Long Head of Biceps Tendon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD 246/2021
Record Dates: First submitted 2023-01-06; First posted 2023-04-18 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-03

CONDITIONS: Rotator Cuff Tears
Keywords: Massive cuff tears; Biceps autograft; Arthroscopic repair partial or complete; Retear; Superior capsular augmentation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic massive Rotator Cuff Tears Repair without using long head of biceps tendon augmentation (Active Comparator): Arthroscopic repair either complete or partial with medialization or not by anchors without using proximal part of long head of biceps tendon) ( single row or double row )(partial or complete anatomical)
  Interventions: Procedure: Arthroscopic massive rotator cuff repair
- Arthroscopic Massive Rotator Cuff Tears Repair With biceps Augmentation (Experimental): • Single or double row repair technique by Rotator Cuff(RC) anchors. Biceps augmentation will be done via release and mobilize the Long Head of Biceps Tendon from bicipital groove. then the proximal part of long head of biceps tendon will be lateralized towards greater tuberosity crossing the gap by passing 1 limb of the RC anchor using suture passer (scorpion or lasso loop) and the other limb of the same anchor was passed through torn cuff. a horizontal limb of distal part biceps tendon was interpositioned between the Rotator Cuff Tears And humeral head, aiding in biological healing and strengthening poor quality rotator cuff tendons
  Interventions: Procedure: Arthroscopic massive rotator cuff repair with superior capsular augmentation using the long head of biceps tendon

INTERVENTIONS:
Procedure: Arthroscopic massive rotator cuff repair — Arthroscopic massive rotator cuff repair without biceps tendon augmentation either partial or complete repair.
  Arms: Arthroscopic massive Rotator Cuff Tears Repair without using long head of biceps tendon augmentation
Procedure: Arthroscopic massive rotator cuff repair with superior capsular augmentation using the long head of biceps tendon — Arthroscopic massive rotator cuff repair with superior capsular augmentation using the long head of biceps tendon .
  Other Names: Superior capsular augmentation using proximal part of the long head of biceps tendon ( LHBT); Biceps tendon autograft technique.
  Arms: Arthroscopic Massive Rotator Cuff Tears Repair With biceps Augmentation

SUMMARY:
The Goal of this clinical trial is to asses the function of arthroscopic repair with or without superior capsular augmentation using biceps tendon .

DETAILED DESCRIPTION:
All patients included in this clinical trial Will be informed by written consent will undergo a one week screening to determine the eligibility for study entry. Patients who meet the eligibility requirements Will be randomised in a single blinded manner ( patients).

ELIGIBILITY:
Inclusion Criteria:

* age 40 to 80 years old
* Patients with massive rotator cuff tear

Exclusion Criteria:

* patients with glenohumeral arthritis
* Acromioclavicular arthritis that requires distal clavicle resection
* Patients with other intra articular pathology like slap lesion
* Neural damage( brachial plexus injury)
* Revision cases

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Functional shoulder constant score (assess the change pre operative and post operative during study period completion) | 1- preoperative 2- six months post operative 3- one year post operative
  Assess the change of Constant score of the patients pre operative and during follow up duration of the study on multiple periods (a multi-item functional scale assessing pain, activity of daily living , range of motion and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively.)
Functional shoulder ases score (assess the change preoperative and postoperative during study period completion ) | 1- preoperative 2- six months post operative 3- one year post operative
  Assess the change in Ases score pre operative and post operative during study completion on multiple periods ( American shoulder and elbow surgeons standardized form)Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.

SECONDARY OUTCOMES:
Shoulder Pain ( assess the change preoperative and postoperative during the study period completion) | 1 pre operative 2 two weeks post operative 3 six months post operative
  Asses the change in the visual analog score ( zero equal no pain and 10 equal severest pain ) pre operative and post operative during study period on different periods

CONTACTS AND LOCATIONS:
Overall Officials: Amr Mo Abdelhady, Professor, Study Chair — Faculty of medicine Ain shams university; Mohamed Ha Sobhy, Professor, Study Director — Faculty of medicine Ain shams university; Ahmed Ha Khater, professor, Study Director — Faculty of medicine Ain shams university; Yahia Mo Haroun, Lecturer, Study Director — Faculty of medicine Ain shams university; Mostafa Ah Mostafa, Principal Investigator — Faculty of medicine Ain shams university
Locations (1):
- Mostafa Ahmed Mohamed Mostafa,MSC, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No